CLINICAL TRIAL: NCT02682823
Title: Tocilizumab Real-Life Human Factors Validation Study
Brief Title: Tocilizumab Real-Life Human Factors (RLHFs) Validation Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: WA29917
Record Dates: First submitted 2016-02-11; First posted 2016-02-15 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Caregivers (Experimental): CGs will perform injection of SC tocilizumab to a subset of participants with RA using the AI-1000 G2 device. Visit 1 (Day 0) will be conducted for administration training, while Visits 2 and 3 (Days 14 and 28) will be conducted for use/performance evaluation.
  Interventions: Device: AI-1000 G2; Drug: Tocilizumab
- Healthcare Professionals (Experimental): HCPs will perform injection of SC tocilizumab to a subset of participants with RA using the AI-1000 G2 device. Because enrolled HCPs are to be professionally qualified to deliver SC injections, no administration training will be provided. Visits 2 and 3 (Days 14 and 28) will be conducted for use/performance evaluation.
  Interventions: Device: AI-1000 G2; Drug: Tocilizumab
- RA Group 1 (Self-Administration) (Experimental): Participants with RA will perform self-injection of SC tocilizumab with the AI-1000 G2 device. Visit 1 (Day 0) will be conducted for administration training, while Visits 2 and 3 (Days 14 and 28) will be conducted for use/performance evaluation.
  Interventions: Device: AI-1000 G2; Drug: Tocilizumab
- RA Group 2 (Administration by CG) (Other): CGs will perform injection of SC tocilizumab to participants with RA using the AI-1000 G2 device. Visit 1 (Day 0) will be conducted for administration training, while Visits 2 and 3 (Days 14 and 28) will be conducted for use/performance evaluation.
  Interventions: Device: AI-1000 G2; Drug: Tocilizumab
- RA Group 3 (Administration by HCP) (Other): HCPs will perform injection of SC tocilizumab to participants with RA using the AI-1000 G2 device. Because enrolled HCPs are to be professionally qualified to deliver SC injections, no administration training will be provided. Visit 1 (Day 0) will be performed by the study nurse. Visits 2 and 3 (Days 14 and 28) will be conducted by the HCP for use/performance evaluation.
  Interventions: Device: AI-1000 G2; Drug: Tocilizumab

INTERVENTIONS:
Device: AI-1000 G2 — Tocilizumab will be administered using the AI-1000 G2.
Drug: Tocilizumab — Participants will receive three doses of SC tocilizumab using the AI-1000 G2 device at Visits 1, 2, and 3 (Days 0, 14, and 28). The dose will remain at 162 milligrams (mg) unless changes are required per protocol for safety or efficacy reasons.
  Other Names: Actemra/RoActemra, RO4877533

SUMMARY:
This study is designed to evaluate RLHFs concerning administration of the tocilizumab autoinjector AI-1000 G2 in adults with rheumatoid arthritis (RA) who have been receiving subcutaneous (SC) tocilizumab using the commercially available prefilled syringe and needle safety device (PFS-NSD). The study will enroll participants with RA, a subset of whom will be assigned to perform self-injection with the AI-1000 G2. Enrolled caregivers (CGs) and healthcare professionals (HCPs) will administer the AI-1000 G2 injection to the remaining study participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants with RA for greater than or equal to (>/=6) months receiving 162 mg tocilizumab PFS-NSD for >/=8 weeks and who are suitable for continued treatment at their currently prescribed dose
* CGs and professionally qualified HCPs who are able and willing to administer the injection

Exclusion Criteria:

* RA: Functional status Class IV
* RA: Neuropathies or other conditions that might interfere with pain evaluation
* RA: Pregnant or breastfeeding
* RA: Low neutrophil or platelet count at last laboratory assessment
* RA: Elevated liver enzymes at last laboratory assessment
* Current participation in another interventional clinical trial
* Criteria that might give the participant/CG/HCP an advantage in injection tasks such as employment in the pharmaceutical industry, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (8):
  - Arizona Arthritis and Rheuma, Mesa, Arizona
  - Valerius Medical Group & Research Ctr of Greater Long Beach, Los Alamitos, California
  - Pacific Arthritis Ctr Med Grp, Santa Maria, California
  - Bluegrass Comm Research, Inc., Lexington, Kentucky
  - Oklahoma Center For Arthritis Therapy & Research, Tulsa, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Advanced Rheumatology & Arthritis Research Center, Wexford, Pennsylvania
  - Metroplex Clinical Research, Dallas, Texas

REFERENCES:
- [Derived] Fettner S, Mela C, Wildenhahn F, Tavanti M, Wells C, Douglass W, Mallalieu NL. Evidence of bioequivalence and positive patient user handling of a tocilizumab autoinjector. Expert Opin Drug Deliv. 2019 May;16(5):551-561. doi: 10.1080/17425247.2019.1604678. Epub 2019 May 2. PMID 31043095

RESULTS

PARTICIPANT FLOW:
Groups:
- Caregivers: Caregivers (CGs) performed injection of 162 milligrams (mg) subcutaneous (SC) tocilizumab to a subset of participants with rheumatoid arthritis (RA) using the AI-1000 G2 device. Visit 1 (Day 0) was conducted for administration training, while Visits 2 and 3 (Days 14 and 28) were conducted for use/performance evaluation.
- Healthcare Professionals: Healthcare professionals (HCPs) performed injection of 162 mg SC tocilizumab to a subset of participants with RA using the AI-1000 G2 device. Because enrolled HCPs were to be professionally qualified to deliver SC injections, no administration training was provided. Visits 2 and 3 (Days 14 and 28) were conducted for use/performance evaluation.
- RA Group 1 (Self-Administration): Participants with RA performed self-injection of 162 mg SC tocilizumab with the AI-1000 G2 device. Visit 1 (Day 0) was conducted for administration training, while Visits 2 and 3 (Days 14 and 28) were conducted for use/performance evaluation.
- RA Group 2 (Administration by CG): CGs performed injection of 162 mg SC tocilizumab to participants with RA using the AI-1000 G2 device. Visit 1 (Day 0) was conducted for administration training, while Visits 2 and 3 (Days 14 and 28) were conducted for use/performance evaluation.
- RA Group 3 (Administration by HCP): HCPs performed injection of 162 mg SC tocilizumab to participants with RA using the AI-1000 G2 device. Because enrolled HCPs were to be professionally qualified to deliver SC injections, no administration training was provided. Visit 1 (Day 0) was performed by the study nurse. Visits 2 and 3 (Days 14 and 28) were conducted by the HCP for use/performance evaluation.
Period: Overall Study
Arm/Group | Caregivers | Healthcare Professionals | RA Group 1 (Self-Administration) | RA Group 2 (Administration by CG) | RA Group 3 (Administration by HCP)
Started | 17 | 19 | 19 | 17 | 19
Safety Population | 17 (All CGs who administered at least one dose of study drug.) | 19 (All HCPs who administered at least one dose of study drug.) | 18 (All participants who received at least one dose of study drug.) | 17 (All participants who received at least one dose of study drug.) | 19 (All participants who received at least one dose of study drug.)
Completed | 17 | 18 | 18 | 16 | 18
Not Completed | 0 | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1
Not completed — Protocol Deviation | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received (or in the case of CGs and HCPs, administered) at least one dose of study drug.
Groups:
- Caregivers: CGs performed injection of 162 mg SC tocilizumab to a subset of participants with RA using the AI-1000 G2 device. Visit 1 (Day 0) was conducted for administration training, while Visits 2 and 3 (Days 14 and 28) were conducted for use/performance evaluation.
- Healthcare Professionals: HCPs performed injection of 162 mg SC tocilizumab to a subset of participants with RA using the AI-1000 G2 device. Because enrolled HCPs were to be professionally qualified to deliver SC injections, no administration training was provided. Visits 2 and 3 (Days 14 and 28) were conducted for use/performance evaluation.
- Total: Total of all reporting groups
Arm/Group | Caregivers | Healthcare Professionals | RA Group 1 (Self-Administration) | RA Group 2 (Administration by CG) | RA Group 3 (Administration by HCP) | Total
Number analyzed (Participants) | 17 | 19 | 18 | 17 | 19 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 14 | 15 | 16 | 77
  >=65 years | 2 | 2 | 4 | 2 | 3 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 13 | 13 | 13 | 68
  Male | 5 | 2 | 5 | 4 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Successfully Performed Safety-Critical and Essential Tasks During First Unassisted Use
Description: Safety-critical tasks included those tasks where errors would have a reasonably foreseeable potential for clinical impact/harm, potentially resulting in direct physical injury to the user and/or conditions that require medical intervention. Safety-critical tasks included the following: release activation button; check the expiry date; inspect device prior to use; and inspect medication prior to use. Essential tasks included those essential to the execution of the injection. Essential tasks included the following: open the carton, remove the device and associated documents; remove cap; start an injection by depressing the needle-shield at the injection site and pressing the activation button; and hold the autoinjector until the complete dose has been delivered. The percentage of participants who successfully performed safety-critical and essential tasks during the first unassisted use (Day 14) was reported.
Time Frame: Day 14
Population: Safety Population; only those who performed the administration task(s) on Day 14 were included because the endpoint was not applicable to non-injecting participants. Here, "n" refers to number evaluable for the specified assessment, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | RA Group 1 (Self-Administration) | Caregivers | Healthcare Professionals
Number analyzed (Participants) | 17 | 17 | 18
percentage of participants
  Open carton, remove device/documents | 100.00 | 100.00 | 100.00
  Remove cap | 100.00 | 100.00 | 100.00
  Start injection: number analyzed (Participants) | 16 | 17 | 18
  Start injection | 93.75 | 94.12 | 100.00
  Hold until complete dose delivered: number analyzed (Participants) | 15 | 16 | 18
  Hold until complete dose delivered | 100.00 | 100.00 | 100.00
  Release activation button: number analyzed (Participants) | 15 | 16 | 18
  Release activation button | 100.00 | 100.00 | 100.00
  Check expiry date | 88.24 | 58.82 | 72.22
  Inspect device prior to use | 76.47 | 47.06 | 66.67
  Inspect medication prior to use | 82.35 | 82.35 | 88.89

2. Primary Outcome: Percentage of Participants Who Successfully Performed Safety-Critical and Essential Tasks During Second Unassisted Use
Description: Safety-critical tasks included those tasks where errors would have a reasonably foreseeable potential for clinical impact/harm, potentially resulting in direct physical injury to the user and/or conditions that require medical intervention. Safety-critical tasks included the following: release activation button; check the expiry date; inspect device prior to use; and inspect medication prior to use. Essential tasks included those essential to the execution of the injection. Essential tasks included the following: open the carton, remove the device and associated documents; remove cap; start an injection by depressing the needle-shield at the injection site and pressing the activation button; and hold the autoinjector until the complete dose has been delivered. The percentage of participants who successfully performed safety-critical and essential tasks during the second unassisted use (Day 28) was reported.
Time Frame: Day 28
Population: Safety Population; only those who performed the administration task(s) on Day 28 were included because the endpoint was not applicable to non-injecting participants.
Measure: Number; unit: percentage of participants
Arm/Group | RA Group 1 (Self-Administration) | Caregivers | Healthcare Professionals
Number analyzed (Participants) | 18 | 17 | 18
percentage of participants
  Open carton, remove device/documents | 100.00 | 100.00 | 100.00
  Remove cap | 100.00 | 100.00 | 100.00
  Start injection | 100.00 | 100.00 | 100.00
  Hold until complete dose delivered | 100.00 | 100.00 | 100.00
  Release activation button | 100.00 | 100.00 | 100.00
  Check expiry date | 94.44 | 76.47 | 94.44
  Inspect device prior to use | 77.78 | 58.82 | 83.33
  Inspect medication prior to use | 88.89 | 70.59 | 94.44

3. Secondary Outcome: Percentage of Participants Who Successfully Performed Ancillary Tasks During First and Second Unassisted Use
Description: Ancillary tasks included those tasks where the potential harm resulting from use error would be minor in severity, or the resultant harms were estimated to occur at sufficiently low levels. Ancillary tasks included the following: wash hands; clean the injection site with alcohol swab; wait for the alcohol to dry; dispose of the autoinjector cap; inspect full dose delivered after use; dispose of the autoinjector; and treatment of injection site after injection. The percentage of participants who succesffully performed ancillary tasks during the first (Day 14) and second unassisted use (Day 28) was reported.
Time Frame: Days 14, 28
Population: Safety Population; only those who performed the administration task(s) were included because the endpoint was not applicable to non-injecting participants. Here, "n" refers to number evaluable for the specified assessment, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | RA Group 1 (Self-Administration) | Caregivers | Healthcare Professionals
Number analyzed (Participants) | 18 | 17 | 18
percentage of participants
  Day (D) 14, wash hands: number analyzed (Participants) | 17 | 17 | 18
  Day (D) 14, wash hands | 82.35 | 82.35 | 77.78
  D28, wash hands | 88.89 | 94.12 | 100.00
  D14, clean/swab injection site: number analyzed (Participants) | 17 | 17 | 18
  D14, clean/swab injection site | 100.00 | 100.00 | 100.00
  D28, clean/swab injection site | 94.44 | 100.00 | 100.00
  D14, wait for alcohol to dry: number analyzed (Participants) | 17 | 17 | 18
  D14, wait for alcohol to dry | 94.12 | 94.12 | 88.89
  D28, wait for alcohol to dry: number analyzed (Participants) | 17 | 17 | 18
  D28, wait for alcohol to dry | 82.35 | 100.00 | 83.33
  D14, dispose of device cap: number analyzed (Participants) | 17 | 15 | 18
  D14, dispose of device cap | 94.12 | 86.67 | 83.33
  D28, dispose of device cap | 94.44 | 88.24 | 94.44
  D14, inspect full dose delivered: number analyzed (Participants) | 15 | 16 | 18
  D14, inspect full dose delivered | 100.00 | 100.00 | 100.00
  D28, inspect full dose delivered | 94.44 | 94.12 | 100.00
  D14, dispose of device: number analyzed (Participants) | 15 | 16 | 18
  D14, dispose of device | 93.33 | 100.00 | 100.00
  D28, dispose of device | 94.44 | 94.12 | 100.00
  D14, treatment of site post injection: number analyzed (Participants) | 15 | 16 | 18
  D14, treatment of site post injection | 100.00 | 100.00 | 100.00
  D28, treatment of site post injection | 100.00 | 100.00 | 100.00

4. Secondary Outcome: Visual Analog Scale (VAS) Score for Injection Pain Among Participants With RA
Description: Injection pain was assessed on a continuous 100-millimeter (mm) VAS, where 0 mm represents "no pain" and 100 mm represents "unbearable pain". The mean VAS response at each assessment timepoint was reported among participants with RA.
Time Frame: 0 and 15 minutes after injection on Days 0, 14, 28
Population: Safety Population; only participants with RA were included because the endpoint was not applicable to CGs and HCPs. Here, "n" refers to number evaluable for the specified assessment, respectively.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Group 1 (Self-Administration) | RA Group 2 (Administration by CG) | RA Group 3 (Administration by HCP)
Number analyzed (Participants) | 18 | 17 | 19
mm
  D0, 0 minutes (min) | 2.8 (4.0) | 9.9 (13.7) | 13.3 (22.9)
  D0, 15min | 1.2 (2.3) | 0.9 (1.9) | 0.8 (1.9)
  D14, 0min: number analyzed (Participants) | 17 | 17 | 17
  D14, 0min | 5.4 (12.9) | 5.0 (7.0) | 11.4 (17.3)
  D14, 15min: number analyzed (Participants) | 17 | 17 | 17
  D14, 15min | 1.5 (2.8) | 0.5 (0.9) | 0.7 (1.4)
  D28, 0min: number analyzed (Participants) | 18 | 16 | 18
  D28, 0min | 4.5 (5.2) | 5.8 (9.0) | 14.5 (20.1)
  D28, 15min: number analyzed (Participants) | 18 | 16 | 18
  D28, 15min | 0.6 (1.5) | 1.9 (5.7) | 0.7 (1.2)

5. Secondary Outcome: Percentage of Participants by Response to Categorical Scale of Injection Pain Among Participants With RA
Description: Injection pain was assessed on a categorical 6-point Likert scale, ranging from "no pain" to "severe and intolerable". The percentage of participants was reported by response at each assessment timepoint among participants with RA.
Time Frame: 0 and 15 minutes after injection on Days 0, 14, 28
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | RA Group 1 (Self-Administration) | RA Group 2 (Administration by CG) | RA Group 3 (Administration by HCP)
Number analyzed (Participants) | 18 | 17 | 19
percentage of participants
  D0, 0min, no pain | 66.7 | 47.1 | 47.4
  D0, 0min, minimal but tolerable | 33.3 | 41.2 | 21.1
  D0, 0min, mild but tolerable | 0 | 11.8 | 21.1
  D0, 0min, moderate but tolerable | 0 | 0 | 5.3
  D0, 0min, moderate-severe/tolerable | 0 | 0 | 5.3
  D0, 0min, severe and intolerable | 0 | 0 | 0
  D0, 15min, no pain | 88.9 | 100.0 | 94.7
  D0, 15min, minimal but tolerable | 11.1 | 0 | 5.3
  D0, 15min, mild but tolerable | 0 | 0 | 0
  D0, 15min, moderate but tolerable | 0 | 0 | 0
  D0, 15min, moderate-severe/tolerable | 0 | 0 | 0
  D0, 15min, severe and intolerable | 0 | 0 | 0
  D14, 0min, no pain: number analyzed (Participants) | 17 | 17 | 17
  D14, 0min, no pain | 70.6 | 64.7 | 52.9
  D14, 0min, minimal but tolerable: number analyzed (Participants) | 17 | 17 | 17
  D14, 0min, minimal but tolerable | 23.5 | 35.3 | 17.6
  D14, 0min, mild but tolerable: number analyzed (Participants) | 17 | 17 | 17
  D14, 0min, mild but tolerable | 5.9 | 0 | 11.8
  D14, 0min, moderate but tolerable: number analyzed (Participants) | 17 | 17 | 17
  D14, 0min, moderate but tolerable | 0 | 0 | 5.9
  D14, 0min, moderate-severe/tolerable: number analyzed (Participants) | 17 | 17 | 17
  D14, 0min, moderate-severe/tolerable | 0 | 0 | 11.8
  D14, 0min, severe and intolerable: number analyzed (Participants) | 17 | 17 | 17
  D14, 0min, severe and intolerable | 0 | 0 | 0
  D14, 15min, no pain: number analyzed (Participants) | 17 | 17 | 17
  D14, 15min, no pain | 88.2 | 100.0 | 82.4
  D14, 15min, minimal but tolerable: number analyzed (Participants) | 17 | 17 | 17
  D14, 15min, minimal but tolerable | 11.8 | 0 | 17.6
  D14, 15min, mild but tolerable: number analyzed (Participants) | 17 | 17 | 17
  D14, 15min, mild but tolerable | 0 | 0 | 0
  D14, 15min, moderate but tolerable: number analyzed (Participants) | 17 | 17 | 17
  D14, 15min, moderate but tolerable | 0 | 0 | 0
  D14, 15min, moderate-severe/tolerable: number analyzed (Participants) | 17 | 17 | 17
  D14, 15min, moderate-severe/tolerable | 0 | 0 | 0
  D14, 15min, severe and intolerable: number analyzed (Participants) | 17 | 17 | 17
  D14, 15min, severe and intolerable | 0 | 0 | 0
  D28, 0min, no pain: number analyzed (Participants) | 18 | 16 | 18
  D28, 0min, no pain | 72.2 | 68.8 | 55.6
  D28, 0min, minimal but tolerable: number analyzed (Participants) | 18 | 16 | 18
  D28, 0min, minimal but tolerable | 27.8 | 18.8 | 33.3
  D28, 0min, mild but tolerable: number analyzed (Participants) | 18 | 16 | 18
  D28, 0min, mild but tolerable | 0 | 12.5 | 5.6
  D28, 0min, moderate but tolerable: number analyzed (Participants) | 18 | 16 | 18
  D28, 0min, moderate but tolerable | 0 | 0 | 5.6
  D28, 0min, moderate-severe/tolerable: number analyzed (Participants) | 18 | 16 | 18
  D28, 0min, moderate-severe/tolerable | 0 | 0 | 0
  D28, 0min, severe and intolerable: number analyzed (Participants) | 18 | 16 | 18
  D28, 0min, severe and intolerable | 0 | 0 | 0
  D28, 15min, no pain: number analyzed (Participants) | 18 | 16 | 18
  D28, 15min, no pain | 100.0 | 100.0 | 88.9
  D28, 15min, minimal but tolerable: number analyzed (Participants) | 18 | 16 | 18
  D28, 15min, minimal but tolerable | 0 | 0 | 11.1
  D28, 15min, mild but tolerable: number analyzed (Participants) | 18 | 16 | 18
  D28, 15min, mild but tolerable | 0 | 0 | 0
  D28, 15min, moderate but tolerable: number analyzed (Participants) | 18 | 16 | 18
  D28, 15min, moderate but tolerable | 0 | 0 | 0
  D28, 15min, moderate-severe/tolerable: number analyzed (Participants) | 18 | 16 | 18
  D28, 15min, moderate-severe/tolerable | 0 | 0 | 0
  D28, 15min, severe and intolerable: number analyzed (Participants) | 18 | 16 | 18
  D28, 15min, severe and intolerable | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants by Response to Device Satisfaction Questionnaire
Description: Device satisfaction was assessed using twelve questions on a categorical 5-point Likert scale, ranging from "strongly agree" to "strongly disagree". Question (Q) 1 (felt the autoinjection was easy to use), Q2 (felt comfortable while using the autoinjector), Q3 (felt the autoinjector was easy to hold), Q4 (able to tell when injection had completed), Q5 (felt he/she can inject properly with the autoinjector), Q6 (felt he/she had control over the injection process), Q7 (felt confident that he/she injected successfully), Q8 (felt it is easy to dispose of the autoinjector), Q9 (autoinjector would help to manage his/her injection schedule), Q10 (liked the look/feel of the autoinjector), Q11 (would recommend the autoinjector to someone else who needed to inject), Q12 (would continue having injections with the autoinjector). The percentage of participants was reported by response at each assessment among participants with RA, CGs, and HCPs.
Time Frame: Days 0, 14, 28
Population: Safety Population. Here, "n" refers to number evaluable for the specified assessment, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | RA Group 1 (Self-Administration) | Caregivers | Healthcare Professionals | RA Group 2 (Administration by CG) | RA Group 3 (Administration by HCP)
Number analyzed (Participants) | 19 | 17 | 19 | 17 | 19
percentage of participants
  Q1, D0, strongly disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q1, D0, strongly disagree | 0 | 0 |  |  |
  Q1, D0, disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q1, D0, disagree | 0 | 0 |  |  |
  Q1, D0, neutral: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q1, D0, neutral | 5.6 | 5.9 |  |  |
  Q1, D0, agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q1, D0, agree | 11.1 | 0 |  |  |
  Q1, D0, strongly agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q1, D0, strongly agree | 83.3 | 94.1 |  |  |
  Q1, D14, strongly disagree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q1, D14, strongly disagree | 11.8 | 6.3 | 0 |  |
  Q1, D14, disagree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q1, D14, disagree | 0 | 0 | 0 |  |
  Q1, D14, neutral: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q1, D14, neutral | 0 | 0 | 5.3 |  |
  Q1, D14, agree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q1, D14, agree | 11.8 | 12.5 | 36.8 |  |
  Q1, D14, strongly agree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q1, D14, strongly agree | 76.5 | 81.3 | 57.9 |  |
  Q1, D28, strongly disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q1, D28, strongly disagree | 0 | 0 | 0 |  |
  Q1, D28, disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q1, D28, disagree | 0 | 11.8 | 0 |  |
  Q1, D28, neutral: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q1, D28, neutral | 0 | 0 | 0 |  |
  Q1, D28, agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q1, D28, agree | 16.7 | 11.8 | 27.8 |  |
  Q1, D28, strongly agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q1, D28, strongly agree | 83.3 | 76.5 | 72.2 |  |
  Q2, D0, strongly disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q2, D0, strongly disagree | 0 | 0 |  |  |
  Q2, D0, disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q2, D0, disagree | 0 | 5.9 |  |  |
  Q2, D0, neutral: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q2, D0, neutral | 0 | 0 |  |  |
  Q2, D0, agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q2, D0, agree | 22.2 | 11.8 |  |  |
  Q2, D0, strongly agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q2, D0, strongly agree | 77.8 | 82.4 |  |  |
  Q2, D14, strongly disagree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q2, D14, strongly disagree | 5.9 | 0 | 0 |  |
  Q2, D14, disagree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q2, D14, disagree | 0 | 6.3 | 0 |  |
  Q2, D14, neutral: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q2, D14, neutral | 0 | 0 | 0 |  |
  Q2, D14, agree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q2, D14, agree | 23.5 | 12.5 | 42.1 |  |
  Q2, D14, strongly agree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q2, D14, strongly agree | 70.6 | 81.3 | 57.9 |  |
  Q2, D28, strongly disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q2, D28, strongly disagree | 0 | 0 | 0 |  |
  Q2, D28, disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q2, D28, disagree | 0 | 11.8 | 0 |  |
  Q2, D28, neutral: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q2, D28, neutral | 0 | 0 | 0 |  |
  Q2, D28, agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q2, D28, agree | 16.7 | 11.8 | 27.8 |  |
  Q2, D28, strongly agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q2, D28, strongly agree | 83.3 | 76.5 | 72.2 |  |
  Q3, D0, strongly disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q3, D0, strongly disagree | 0 | 0 |  |  |
  Q3, D0, disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q3, D0, disagree | 5.6 | 0 |  |  |
  Q3, D0, neutral: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q3, D0, neutral | 5.6 | 5.9 |  |  |
  Q3, D0, agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q3, D0, agree | 27.8 | 5.9 |  |  |
  Q3, D0, strongly agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q3, D0, strongly agree | 61.1 | 88.2 |  |  |
  Q3, D14, strongly disagree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q3, D14, strongly disagree | 5.9 | 0 | 0 |  |
  Q3, D14, disagree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q3, D14, disagree | 5.9 | 6.3 | 0 |  |
  Q3, D14, neutral: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q3, D14, neutral | 0 | 6.3 | 0 |  |
  Q3, D14, agree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q3, D14, agree | 17.6 | 18.8 | 31.6 |  |
  Q3, D14, strongly agree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q3, D14, strongly agree | 70.6 | 68.8 | 68.4 |  |
  Q3, D28, strongly disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q3, D28, strongly disagree | 0 | 0 | 0 |  |
  Q3, D28, disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q3, D28, disagree | 0 | 5.9 | 0 |  |
  Q3, D28, neutral: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q3, D28, neutral | 0 | 0 | 0 |  |
  Q3, D28, agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q3, D28, agree | 16.7 | 11.8 | 22.2 |  |
  Q3, D28, strongly agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q3, D28, strongly agree | 83.3 | 82.4 | 77.8 |  |
  Q4, D0, strongly disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q4, D0, strongly disagree | 0 | 0 |  |  |
  Q4, D0, disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q4, D0, disagree | 11.1 | 5.9 |  |  |
  Q4, D0, neutral: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q4, D0, neutral | 0 | 5.9 |  |  |
  Q4, D0, agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q4, D0, agree | 44.4 | 17.6 |  |  |
  Q4, D0, strongly agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q4, D0, strongly agree | 44.4 | 70.6 |  |  |
  Q4, D14, strongly disagree: number analyzed (Participants) | 17 | 15 | 19 | 0 | 0
  Q4, D14, strongly disagree | 5.9 | 0 | 0 |  |
  Q4, D14, disagree: number analyzed (Participants) | 17 | 15 | 19 | 0 | 0
  Q4, D14, disagree | 5.9 | 6.7 | 0 |  |
  Q4, D14, neutral: number analyzed (Participants) | 17 | 15 | 19 | 0 | 0
  Q4, D14, neutral | 11.8 | 0 | 0 |  |
  Q4, D14, agree: number analyzed (Participants) | 17 | 15 | 19 | 0 | 0
  Q4, D14, agree | 17.6 | 13.3 | 31.6 |  |
  Q4, D14, strongly agree: number analyzed (Participants) | 17 | 15 | 19 | 0 | 0
  Q4, D14, strongly agree | 58.8 | 80.0 | 68.4 |  |
  Q4, D28, strongly disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q4, D28, strongly disagree | 0 | 5.9 | 0 |  |
  Q4, D28, disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q4, D28, disagree | 0 | 0 | 0 |  |
  Q4, D28, neutral: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q4, D28, neutral | 0 | 0 | 0 |  |
  Q4, D28, agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q4, D28, agree | 22.2 | 11.8 | 16.7 |  |
  Q4, D28, strongly agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q4, D28, strongly agree | 77.8 | 82.4 | 83.3 |  |
  Q5, D0, strongly disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q5, D0, strongly disagree | 0 | 0 |  |  |
  Q5, D0, disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q5, D0, disagree | 0 | 0 |  |  |
  Q5, D0, neutral: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q5, D0, neutral | 11.1 | 0 |  |  |
  Q5, D0, agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q5, D0, agree | 22.2 | 11.8 |  |  |
  Q5, D0, strongly agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q5, D0, strongly agree | 66.7 | 88.2 |  |  |
  Q5, D14, strongly disagree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q5, D14, strongly disagree | 5.9 | 0 | 0 |  |
  Q5, D14, disagree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q5, D14, disagree | 0 | 6.3 | 0 |  |
  Q5, D14, neutral: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q5, D14, neutral | 5.9 | 6.3 | 0 |  |
  Q5, D14, agree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q5, D14, agree | 11.8 | 0 | 15.8 |  |
  Q5, D14, strongly agree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q5, D14, strongly agree | 76.5 | 87.5 | 84.2 |  |
  Q5, D28, strongly disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q5, D28, strongly disagree | 0 | 0 | 0 |  |
  Q5, D28, disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q5, D28, disagree | 0 | 5.9 | 0 |  |
  Q5, D28, neutral: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q5, D28, neutral | 0 | 0 | 0 |  |
  Q5, D28, agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q5, D28, agree | 16.7 | 11.8 | 22.2 |  |
  Q5, D28, strongly agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q5, D28, strongly agree | 83.3 | 82.4 | 77.8 |  |
  Q6, D0, strongly disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q6, D0, strongly disagree | 0 | 0 |  |  |
  Q6, D0, disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q6, D0, disagree | 5.6 | 0 |  |  |
  Q6, D0, neutral: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q6, D0, neutral | 5.6 | 5.9 |  |  |
  Q6, D0, agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q6, D0, agree | 16.7 | 5.9 |  |  |
  Q6, D0, strongly agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q6, D0, strongly agree | 72.2 | 88.2 |  |  |
  Q6, D14, strongly disagree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q6, D14, strongly disagree | 5.9 | 0 | 0 |  |
  Q6, D14, disagree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q6, D14, disagree | 5.9 | 6.3 | 0 |  |
  Q6, D14, neutral: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q6, D14, neutral | 0 | 6.3 | 0 |  |
  Q6, D14, agree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q6, D14, agree | 11.8 | 12.5 | 26.3 |  |
  Q6, D14, strongly agree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q6, D14, strongly agree | 76.5 | 75.0 | 73.7 |  |
  Q6, D28, strongly disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q6, D28, strongly disagree | 0 | 0 | 0 |  |
  Q6, D28, disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q6, D28, disagree | 0 | 0 | 0 |  |
  Q6, D28, neutral: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q6, D28, neutral | 0 | 5.9 | 0 |  |
  Q6, D28, agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q6, D28, agree | 16.7 | 11.8 | 22.2 |  |
  Q6, D28, strongly agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q6, D28, strongly agree | 83.3 | 82.4 | 77.8 |  |
  Q7, D0, strongly disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q7, D0, strongly disagree | 0 | 0 |  |  |
  Q7, D0, disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q7, D0, disagree | 11.1 | 5.9 |  |  |
  Q7, D0, neutral: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q7, D0, neutral | 0 | 0 |  |  |
  Q7, D0, agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q7, D0, agree | 16.7 | 17.6 |  |  |
  Q7, D0, strongly agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q7, D0, strongly agree | 72.2 | 76.5 |  |  |
  Q7, D14, strongly disagree: number analyzed (Participants) | 17 | 15 | 19 | 0 | 0
  Q7, D14, strongly disagree | 5.9 | 0 | 0 |  |
  Q7, D14, disagree: number analyzed (Participants) | 17 | 15 | 19 | 0 | 0
  Q7, D14, disagree | 0 | 0 | 0 |  |
  Q7, D14, neutral: number analyzed (Participants) | 17 | 15 | 19 | 0 | 0
  Q7, D14, neutral | 5.9 | 0 | 0 |  |
  Q7, D14, agree: number analyzed (Participants) | 17 | 15 | 19 | 0 | 0
  Q7, D14, agree | 17.6 | 6.7 | 21.1 |  |
  Q7, D14, strongly agree: number analyzed (Participants) | 17 | 15 | 19 | 0 | 0
  Q7, D14, strongly agree | 70.6 | 93.3 | 78.9 |  |
  Q7, D28, strongly disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q7, D28, strongly disagree | 0 | 5.9 | 0 |  |
  Q7, D28, disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q7, D28, disagree | 0 | 0 | 0 |  |
  Q7, D28, neutral: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q7, D28, neutral | 0 | 0 | 0 |  |
  Q7, D28, agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q7, D28, agree | 16.7 | 11.8 | 11.1 |  |
  Q7, D28, strongly agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q7, D28, strongly agree | 83.3 | 82.4 | 88.9 |  |
  Q8, D0, strongly disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q8, D0, strongly disagree | 0 | 0 |  |  |
  Q8, D0, disagree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q8, D0, disagree | 0 | 0 |  |  |
  Q8, D0, neutral: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q8, D0, neutral | 0 | 0 |  |  |
  Q8, D0, agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q8, D0, agree | 16.7 | 5.9 |  |  |
  Q8, D0, strongly agree: number analyzed (Participants) | 18 | 17 | 0 | 0 | 0
  Q8, D0, strongly agree | 83.3 | 94.1 |  |  |
  Q8, D14, strongly disagree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q8, D14, strongly disagree | 0 | 0 | 0 |  |
  Q8, D14, disagree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q8, D14, disagree | 5.9 | 0 | 0 |  |
  Q8, D14, neutral: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q8, D14, neutral | 0 | 0 | 0 |  |
  Q8, D14, agree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q8, D14, agree | 17.6 | 0 | 10.5 |  |
  Q8, D14, strongly agree: number analyzed (Participants) | 17 | 16 | 19 | 0 | 0
  Q8, D14, strongly agree | 76.5 | 100.0 | 89.5 |  |
  Q8, D28, strongly disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q8, D28, strongly disagree | 0 | 0 | 0 |  |
  Q8, D28, disagree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q8, D28, disagree | 0 | 5.9 | 0 |  |
  Q8, D28, neutral: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q8, D28, neutral | 0 | 0 | 0 |  |
  Q8, D28, agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q8, D28, agree | 16.7 | 11.8 | 11.1 |  |
  Q8, D28, strongly agree: number analyzed (Participants) | 18 | 17 | 18 | 0 | 0
  Q8, D28, strongly agree | 83.3 | 82.4 | 88.9 |  |
  Q9, D0, strongly disagree: number analyzed (Participants) | 18 | 0 | 0 | 14 | 17
  Q9, D0, strongly disagree | 0 |  |  | 7.1 | 0
  Q9, D0, disagree: number analyzed (Participants) | 18 | 0 | 0 | 14 | 17
  Q9, D0, disagree | 0 |  |  | 0 | 0
  Q9, D0, neutral: number analyzed (Participants) | 18 | 0 | 0 | 14 | 17
  Q9, D0, neutral | 5.6 |  |  | 7.1 | 17.6
  Q9, D0, agree: number analyzed (Participants) | 18 | 0 | 0 | 14 | 17
  Q9, D0, agree | 38.9 |  |  | 28.6 | 29.4
  Q9, D0, strongly agree: number analyzed (Participants) | 18 | 0 | 0 | 14 | 17
  Q9, D0, strongly agree | 55.6 |  |  | 57.1 | 52.9
  Q9, D14, strongly disagree: number analyzed (Participants) | 17 | 0 | 0 | 16 | 17
  Q9, D14, strongly disagree | 0 |  |  | 0 | 0
  Q9, D14, disagree (n=17,0,0,16,17): number analyzed (Participants) | 17 | 0 | 0 | 16 | 17
  Q9, D14, disagree (n=17,0,0,16,17) | 0 |  |  | 0 | 0
  Q9, D14, neutral: number analyzed (Participants) | 17 | 0 | 0 | 16 | 17
  Q9, D14, neutral | 5.9 |  |  | 12.5 | 23.5
  Q9, D14, agree: number analyzed (Participants) | 17 | 0 | 0 | 16 | 17
  Q9, D14, agree | 35.3 |  |  | 18.8 | 23.5
  Q9, D14, strongly agree: number analyzed (Participants) | 17 | 0 | 0 | 16 | 17
  Q9, D14, strongly agree | 58.8 |  |  | 68.8 | 52.9
  Q9, D28, strongly disagree: number analyzed (Participants) | 18 | 0 | 0 | 16 | 18
  Q9, D28, strongly disagree | 0 |  |  | 0 | 5.6
  Q9, D28, disagree: number analyzed (Participants) | 18 | 0 | 0 | 16 | 18
  Q9, D28, disagree | 0 |  |  | 0 | 0
  Q9, D28, neutral: number analyzed (Participants) | 18 | 0 | 0 | 16 | 18
  Q9, D28, neutral | 0 |  |  | 12.5 | 16.7
  Q9, D28, agree: number analyzed (Participants) | 18 | 0 | 0 | 16 | 18
  Q9, D28, agree | 27.8 |  |  | 18.8 | 33.3
  Q9, D28, strongly agree: number analyzed (Participants) | 18 | 0 | 0 | 16 | 18
  Q9, D28, strongly agree | 72.2 |  |  | 68.8 | 44.4
  Q10, D0, strongly disagree: number analyzed (Participants) | 18 | 17 | 0 | 14 | 17
  Q10, D0, strongly disagree | 0 | 0 |  | 7.1 | 0
  Q10, D0, disagree: number analyzed (Participants) | 18 | 17 | 0 | 14 | 17
  Q10, D0, disagree | 0 | 0 |  | 0 | 0
  Q10, D0, neutral: number analyzed (Participants) | 18 | 17 | 0 | 14 | 17
  Q10, D0, neutral | 11.1 | 11.8 |  | 7.1 | 11.8
  Q10, D0, agree: number analyzed (Participants) | 18 | 17 | 0 | 14 | 17
  Q10, D0, agree | 33.3 | 11.8 |  | 21.4 | 41.2
  Q10, D0, strongly agree: number analyzed (Participants) | 18 | 17 | 0 | 14 | 17
  Q10, D0, strongly agree | 55.6 | 76.5 |  | 64.3 | 47.1
  Q10, D14, strongly disagree: number analyzed (Participants) | 17 | 16 | 19 | 16 | 17
  Q10, D14, strongly disagree | 5.9 | 0 | 0 | 0 | 0
  Q10, D14, disagree: number analyzed (Participants) | 17 | 16 | 19 | 16 | 17
  Q10, D14, disagree | 5.9 | 0 | 0 | 6.3 | 5.9
  Q10, D14, neutral: number analyzed (Participants) | 17 | 16 | 19 | 16 | 17
  Q10, D14, neutral | 0 | 0 | 0 | 6.3 | 11.8
  Q10, D14, agree: number analyzed (Participants) | 17 | 16 | 19 | 16 | 17
  Q10, D14, agree | 23.5 | 43.8 | 31.6 | 12.5 | 41.2
  Q10, D14, strongly agree: number analyzed (Participants) | 17 | 16 | 19 | 16 | 17
  Q10, D14, strongly agree | 64.7 | 56.3 | 68.4 | 75.0 | 41.2
  Q10, D28, strongly disagree: number analyzed (Participants) | 18 | 17 | 18 | 16 | 18
  Q10, D28, strongly disagree | 0 | 5.9 | 0 | 0 | 0
  Q10, D28, disagree: number analyzed (Participants) | 18 | 17 | 18 | 16 | 18
  Q10, D28, disagree | 0 | 0 | 0 | 0 | 5.6
  Q10, D28, neutral: number analyzed (Participants) | 18 | 17 | 18 | 16 | 18
  Q10, D28, neutral | 11.1 | 0 | 5.6 | 12.5 | 0
  Q10, D28, agree: number analyzed (Participants) | 18 | 17 | 18 | 16 | 18
  Q10, D28, agree | 16.7 | 35.3 | 27.8 | 18.8 | 44.4
  Q10, D28, strongly agree: number analyzed (Participants) | 18 | 17 | 18 | 16 | 18
  Q10, D28, strongly agree | 72.2 | 58.8 | 66.7 | 68.8 | 50.0
  Q11, D0, strongly disagree: number analyzed (Participants) | 18 | 17 | 0 | 14 | 17
  Q11, D0, strongly disagree | 0 | 0 |  | 14.3 | 0
  Q11, D0, disagree: number analyzed (Participants) | 18 | 17 | 0 | 14 | 17
  Q11, D0, disagree | 0 | 0 |  | 0 | 0
  Q11, D0, neutral: number analyzed (Participants) | 18 | 17 | 0 | 14 | 17
  Q11, D0, neutral | 0 | 5.9 |  | 7.1 | 5.9
  Q11, D0, agree: number analyzed (Participants) | 18 | 17 | 0 | 14 | 17
  Q11, D0, agree | 27.8 | 5.9 |  | 21.4 | 35.3
  Q11, D0, strongly agree: number analyzed (Participants) | 18 | 17 | 0 | 14 | 17
  Q11, D0, strongly agree | 72.2 | 88.2 |  | 57.1 | 58.8
  Q11, D14, strongly disagree: number analyzed (Participants) | 17 | 16 | 19 | 16 | 17
  Q11, D14, strongly disagree | 5.9 | 0 | 0 | 0 | 0
  Q11, D14, disagree: number analyzed (Participants) | 17 | 16 | 19 | 16 | 17
  Q11, D14, disagree | 5.9 | 6.3 | 0 | 0 | 0
  Q11, D14, neutral: number analyzed (Participants) | 17 | 16 | 19 | 16 | 17
  Q11, D14, neutral | 0 | 0 | 0 | 6.3 | 11.8
  Q11, D14, agree: number analyzed (Participants) | 17 | 16 | 19 | 16 | 17
  Q11, D14, agree | 11.8 | 18.8 | 21.1 | 12.5 | 35.3
  Q11, D14, strongly agree: number analyzed (Participants) | 17 | 16 | 19 | 16 | 17
  Q11, D14, strongly agree | 76.5 | 75.0 | 78.9 | 81.3 | 52.9
  Q11, D28, strongly disagree: number analyzed (Participants) | 18 | 17 | 18 | 16 | 18
  Q11, D28, strongly disagree | 0 | 5.9 | 0 | 0 | 0
  Q11, D28, disagree: number analyzed (Participants) | 18 | 17 | 18 | 16 | 18
  Q11, D28, disagree | 0 | 5.9 | 0 | 0 | 5.6
  Q11, D28, neutral: number analyzed (Participants) | 18 | 17 | 18 | 16 | 18
  Q11, D28, neutral | 0 | 0 | 0 | 12.5 | 5.6
  Q11, D28, agree: number analyzed (Participants) | 18 | 17 | 18 | 16 | 18
  Q11, D28, agree | 16.7 | 5.9 | 33.3 | 6.3 | 33.3
  Q11, D28, strongly agree: number analyzed (Participants) | 18 | 17 | 18 | 16 | 18
  Q11, D28, strongly agree | 83.3 | 82.4 | 66.7 | 81.3 | 55.6
  Q12, D0, strongly disagree: number analyzed (Participants) | 18 | 0 | 0 | 14 | 17
  Q12, D0, strongly disagree | 0 |  |  | 14.3 | 0
  Q12, D0, disagree: number analyzed (Participants) | 18 | 0 | 0 | 14 | 17
  Q12, D0, disagree | 0 |  |  | 0 | 0
  Q12, D0, neutral: number analyzed (Participants) | 18 | 0 | 0 | 14 | 17
  Q12, D0, neutral | 5.6 |  |  | 0 | 5.9
  Q12, D0, agree: number analyzed (Participants) | 18 | 0 | 0 | 14 | 17
  Q12, D0, agree | 27.8 |  |  | 21.4 | 35.3
  Q12, D0, strongly agree: number analyzed (Participants) | 18 | 0 | 0 | 14 | 17
  Q12, D0, strongly agree | 66.7 |  |  | 64.3 | 58.8
  Q12, D14, strongly disagree: number analyzed (Participants) | 17 | 0 | 0 | 16 | 17
  Q12, D14, strongly disagree | 5.9 |  |  | 0 | 0
  Q12, D14, disagree: number analyzed (Participants) | 17 | 0 | 0 | 16 | 17
  Q12, D14, disagree | 5.9 |  |  | 0 | 5.9
  Q12, D14, neutral: number analyzed (Participants) | 17 | 0 | 0 | 16 | 17
  Q12, D14, neutral | 0 |  |  | 6.3 | 5.9
  Q12, D14, agree: number analyzed (Participants) | 17 | 0 | 0 | 16 | 17
  Q12, D14, agree | 5.9 |  |  | 12.5 | 35.3
  Q12, D14, strongly agree: number analyzed (Participants) | 17 | 0 | 0 | 16 | 17
  Q12, D14, strongly agree | 82.4 |  |  | 81.3 | 52.9
  Q12, D28, strongly disagree: number analyzed (Participants) | 18 | 0 | 0 | 16 | 18
  Q12, D28, strongly disagree | 0 |  |  | 0 | 0
  Q12, D28, disagree: number analyzed (Participants) | 18 | 0 | 0 | 16 | 18
  Q12, D28, disagree | 0 |  |  | 6.3 | 5.6
  Q12, D28, neutral: number analyzed (Participants) | 18 | 0 | 0 | 16 | 18
  Q12, D28, neutral | 5.6 |  |  | 0 | 5.6
  Q12, D28, agree: number analyzed (Participants) | 18 | 0 | 0 | 16 | 18
  Q12, D28, agree | 11.1 |  |  | 25.0 | 33.3
  Q12, D28, strongly agree: number analyzed (Participants) | 18 | 0 | 0 | 16 | 18
  Q12, D28, strongly agree | 83.3 |  |  | 68.8 | 55.6

7. Secondary Outcome: Tender Joint Count (TJC) Among Participants With RA
Description: Sixty-eight joints were assessed for tenderness among participants with RA. The number of tender joints at Baseline was reported.
Time Frame: Baseline (Day 0)
Population: Safety Population; only participants with RA were included because the endpoint was not applicable to CGs and HCPs.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | RA Group 1 (Self-Administration) | RA Group 2 (Administration by CG) | RA Group 3 (Administration by HCP)
Number analyzed (Participants) | 18 | 17 | 19
tender joints | 11.17 (9.32) | 8.12 (11.29) | 16.32 (16.17)

8. Secondary Outcome: Swollen Joint Count (SJC) Among Participants With RA
Description: Sixty-six joints were assessed for swelling among participants with RA. The number of swollen joints at Baseline was reported.
Time Frame: Baseline (Day 0)
Population: Safety Population; only participants with RA were included because the endpoint was not applicable to CGs and HCPs.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | RA Group 1 (Self-Administration) | RA Group 2 (Administration by CG) | RA Group 3 (Administration by HCP)
Number analyzed (Participants) | 18 | 17 | 19
swollen joints | 4.61 (4.10) | 3.71 (4.45) | 8.89 (7.88)

9. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Among Participants With RA
Description: Ability to perform daily living activities was assessed across eight component sets including dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common activities. Twenty questions were scored on a 4-point Likert scale from 0 meaning "without any difficulty" to 3 meaning "unable to do". The overall score was computed as the sum of domain scores divided by the number of domains answered. Therefore, the score range for HAQ-DI was the same as that of the individual questions, that is, from 0 to 3, where 0 indicates "least difficulty" and 3 indicates "extreme difficulty". The mean change from baseline in HAQ-DI at each assessment was reported among participants with RA.
Time Frame: Days 0, 14, 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Group 1 (Self-Administration) | RA Group 2 (Administration by CG) | RA Group 3 (Administration by HCP)
Number analyzed (Participants) | 18 | 17 | 19
units on a scale
  D0 | 0.7222 (0.6974) | 0.8676 (0.6532) | 1.2434 (0.6541)
  Change at D14: number analyzed (Participants) | 18 | 17 | 17
  Change at D14 | 0.0962 (0.2166) | -0.0368 (0.1863) | -0.0441 (0.2575)
  Change at D28: number analyzed (Participants) | 18 | 16 | 18
  Change at D28 | 0.0139 (0.2674) | -0.0078 (0.2519) | -0.0903 (0.3398)

ADVERSE EVENTS:
Time Frame: Days 0-28
Description: Safety Population; only participants with RA were assessed for adverse events. CGs and HCPs were not included in the analysis.
Arm/Group | RA Group 1 (Self-Administration) | RA Group 2 (Administration by CG) | RA Group 3 (Administration by HCP)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 4/18 | 4/17 | 3/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RA Group 1 (Self-Administration) (N=18) | RA Group 2 (Administration by CG) (N=17) | RA Group 3 (Administration by HCP) (N=19)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/ or the publication be postponed in order to protect the Sponsor's intellectual property rights.